CLINICAL TRIAL: NCT01380002
Title: Home-Care Needs in Liver or Renal Transplantation Recipients and Their Spouses
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Shiow-Ching Shun, NTU
Other Study IDs: 201011063RC
Record Dates: First submitted 2011-06-22; First posted 2011-06-23 (Estimated); Last update posted 2011-06-23 (Estimated); Status verified 2011-06

CONDITIONS: Liver Transplant; Renal Transplant
Keywords: care needs

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

SUMMARY:
* Liver/renal transplantations are now tending to be the most important treatment for terminal liver and renal disease. Although transplantation can prevent recipients from suffering with critical and fatal symptoms, patients may experience the complication from surgery and immunosuppressive drugs. Furthermore, they might have many unmet needs in daily life, and so as their spouses. The purpose of this study is to explore the home-care needs among the post liver or renal transplant recipients and their spouses, and identify the significant factors for care needs.
* A cross-sectional correlated design will be used and patients will be recruited by purposive sampling from an organ transplant outpatient department at a medical center in northern Taiwan. A set of structured questionnaires will be used to collect data.
* The result of this study will be helpful for clinical nurses to understand liver or renal recipients' physical and mental distress, also identify the potential risk of home-care needs and the degree of satisfaction as well.

ELIGIBILITY:
Inclusion Criteria:

* about patients

  1. liver transplant recipients or renal transplant recipients who have regular follow up in organ transplant outpatient departments.
  2. conscious clear.
  3. above 18 years old.
* about spouse

  1. who live with patients.
  2. conscious clear.
  3. above 18 years old.

Exclusion Criteria:

* about patients

  1. who suffer form cancer now.
  2. have received transplantation twice.
* about spouse

  1. who liver apart from patients.
  2. whose spouse(patient) did not recruited in this research.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * liver transplant recipients or renal transplant recipients with 18 to 80 years old who have regular follow up in organ transplant outpatient departments at National Taiwan University Hospital in Northern Taiwan.
  * We will also recuit spouses who live with recruited patients.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2010-12; Primary Completion 2011-10 (Estimated); Study Completion 2011-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Shiow-Ching Shun, Doctor, Study Chair — Department of Nursing
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan